CLINICAL TRIAL: NCT05626712
Title: Clinical Trial to Evaluate the Safety and Efficacy of CELZ-201 in Patients With Recent Onset Type 1 Diabetes (CREATE-1)
Brief Title: Safety and Efficacy of CELZ-201 in Patients With Recent Onset Type 1 Diabetes
Acronym: CREATE-1
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Creative Medical Technology Holdings Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CELZ-201-001
Record Dates: First submitted 2022-11-07; First posted 2022-11-25 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Type 1 Diabetes; Diabetes Mellitus, Type 1
Keywords: Recent Onset Type 1 Diabetes; Adult Onset Type 1 Diabetes; Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: The study is a two-arm, open label, randomized trial. Subjects who meet eligibility criteria will be randomized to treatment or control groups in a 2:1 ratio.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- CELZ-201 Treatment Group (Experimental): Participants in this group will receive a single dose of CELZ-201, in addition to standard of care of care for Type 1 Diabetes treatment.
  Interventions: Biological: CELZ-201 Administration
- Control Group (Placebo Comparator): Participants in this group will receive standard of care for Type 1 Diabetes only.
  Interventions: Other: Control Group

INTERVENTIONS:
Biological: CELZ-201 Administration — Participants in this group will receive a single dose of CELZ-201, in addition to standard of care for Type 1 Diabetes treatment. Perinatal tissue derived cells will be administered at a dose of 1x10^6 cells/kg via an intra-arterial infusion into the dorsal pancreatic artery.
  Arms: CELZ-201 Treatment Group
Other: Control Group — Enhanced standard of care for Type 1 Diabetes treatment only.
  Arms: Control Group

SUMMARY:
The brief purpose of this research study is to learn about the safety and efficacy of intra-arterial administration of CELZ-201 in patients with newly diagnosed Type 1 Diabetes Mellitus (T1D).

DETAILED DESCRIPTION:
The proposed study is a Phase I/IIa randomized, controlled clinical trial to evaluate CELZ-201 therapy as an intervention for the treatment of recent onset Type 1 Diabetes. The objective is to determine the safety and efficacy of CELZ-201 administration, based on the timing and dose of CELZ-201 treatment. Subjects who meet eligibility criteria will be randomized to treatment or control groups, in a 2:1 ratio. Subjects in the Group I (Treatment Group, n=12) will receive standard of care for type 1 diabetes and CELZ-201 within 1 month from enrollment (within 1 year of diagnosis). Subjects in Group II (Control Arm, n=6) and will receive enhanced standard of care for type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be able to understand and provide signed informed consent.
2. Males and females, 18-35 years of age.
3. Diagnosis of T1D within 1 year, with stimulated C-peptide peak level >0.6 ng/mL as assessed by 4-hour MMTT at the time of Visit 0 (screening).
4. Diagnosed with T1D, according to ADA standard criteria, and confirmed by positivity to at least two islet autoantibodies, GAD65, IA-2, or ZnT8.
5. Mentally stable and able to comply with the procedures of the study protocol
6. Subjects must be willing to comply with "standard-of-care" diabetes management.
7. Subjects with eGFR >80 ml/min/1.73m2
8. Female subjects of childbearing potential must have a negative pregnancy test upon study entry.
9. Female (and male) subjects with reproductive potential must agree to use two FDA approved methods of birth control for the entire duration of the study.

   Potential subjects of childbearing potential should agree to use effective contraception for the entire 2-year period.
10. Adequate venous access to support study required blood draws.

Exclusion Criteria:

1. Inability or unwillingness of a subject to give written informed consent or comply with study protocol.
2. BMI>28 kg/m.
3. HbA1c > 9%
4. Subjects with poorly controlled hypertension as defined by systolic blood pressure >140 mmHg or diastolic blood pressure >90 mmHg.
5. Subjects with any history of cardiac disease, including but not limited to myocardial infarction, uncompensated heart failure, fluid overload, as well as any clinically significant abnormality identified on prior cardiac stress test, angiogram evaluation, or echocardiogram.
6. Subjects with liver disease, portal hypertension, any coagulopathy (including history of Factor V deficiency) or long-term anti-coagulant therapy (except low-dose aspirin). Other hepatic conditions including hepatic anatomic abnormalities or variants that would place the individual at increased risk in the judgment of the investigator are also considered exclusionary.
7. Symptomatic cholecystolithiasis; acute or chronic pancreatitis; or current symptomatic peptic ulcer disease.
8. Subjects with uncontrolled thyroid disease: thyroid stimulating hormone <0.3 mU/L or >5 mU/L; free T4 <5.0 ug/dL or >11.0 ug/dL.
9. Any of the following laboratory findings: hemoglobin <11.5 g/dL (females) or <13.2 g/dL (males); leukocytes <3,000/μL; neutrophils <1,500/μL; lymphocytes <800/μL; platelets <100,000/μL; elevation in AST and ALT >2 x ULN (upper limit of normal); LDL cholesterol >160; Triglycerides >3 x ULN; total bilirubin >1.5 x ULN.
10. Screening laboratory evidence consistent with significant chronic active infection (i.e.., hepatitis B and C, tuberculosis, and HIV), and IGRA Tuberculosis (Tb) test during screening
11. Ongoing acute infections, e.g., acute respiratory tract, urinary tract, or gastrointestinal tract infections.
12. Subjects with eating disorders.
13. Ongoing or anticipated use of diabetes medications other than insulin.
14. Current or ongoing use of non-insulin pharmaceuticals that affect glycemic control within 7 days of screening.
15. Recent recipient of any licensed or investigational live attenuated vaccine(s) within 6 weeks of randomization.
16. Patients who have participated in previous clinical studies, other than observational studies, will be excluded.
17. Concomitant therapy with immunosuppressive drugs, immunomodulators, or cytotoxic agents, or previous therapy less than 3 months from randomization.
18. History or diagnosis of malignancy with the exception of a history of localized basal or squamous cell carcinoma.
19. Any history of gastroparesis or other severe gastrointestinal disease.
20. Presence of an allograft.
21. Diagnosed or self-reported drug or alcohol abuse.
22. An individual who has a medical, psychological or social condition that, in the opinion of the Principal Investigator, would interfere with safe and proper completion of the trial.
23. Pregnancy or ongoing breastfeeding for women; unwillingness or inability of both females and males of childbearing age to use a reliable and effective form of contraception, for the entire 2-year duration of the study.
24. Inability to perform any of the assessments required for endpoint analysis.
25. Known history of serious allergic reactions, including anaphylaxis to CELZ-201 or its preparation components. Specifically, patients with a prior history of heparin induced thrombocytopenia or any other adverse reaction to heparin, will be excluded.
26. The investigator believes that participating in the trial is not in the best interest of the patient, or the investigator considers patient unsuitable for enrollment (such as unpredictable risks or subject compliance issues).
27. Positive for coronavirus disease (COVID)-19 by PCR or evidence of active infection per local institutional standards.
28. Allergy to iodine contrast or anesthesia
29. For female subjects: Pregnant, nursing, or planning to become pregnant during the course of entire duration of the study (approximately little over two years) or unwillingness to comply with contraceptive requirements.
30. For male subjects: Male subjects with a female partner who is planning to become pregnant with the male subject during the entire course of the study or unwillingness to comply with contraceptive requirements.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2023-04-07 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events | 6 months
  The primary outcome to be assessed is tolerability and safety of the CELZ-201 therapy. The incidence of adverse events (grade 2 or above as per CTCAE version 5.0) in both groups at 6 months.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events | 12 months
  Incidence of adverse events (grade 2 or above as per CTCAE version 5.0) in both groups at 12 months.
Number of Participants with Adverse Events | 24 months
  Incidence of adverse events (grade 2 or above as per CTCAE version 5.0) in both groups at 24 months.
Glycosylated HbA1C | 12 months
  Changes in glycosylated HbA1c (%)
Insulin Requirement | 12 months
  Changes in exogenous insulin requirement
Islet Autoantibody Levels | 12 months
  Changes in islet autoantibody levels GAD65 (U/mL), IA2 (U/mL), and ZnT8 (U/mL)
Alloreactive Antibody Levels | 12 months
  Changes in alloreactive antibody levels (U/mL)
C-peptide during a 4-hour MMTT | 12 months
  Changes in fasting, peak stimulated and AUC C-peptide (ng/mL) during a 4-hour MMTT

CONTACTS AND LOCATIONS:
Overall Officials: Camillo Ricordi, MD, Principal Investigator — University of Miami, Diabetes Research Institute
Locations (1):
- Diabetes Research Institute, University of Miami Miller School of Medicine, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No